CLINICAL TRIAL: NCT07016867
Title: Medical Treatment Alone Versus Varicocelectomy Versus Varicocelectomy and Medical Treatment in Management of Male Subfertility With Isolated Teratozoospermia: A Prospective Randomized Study
Brief Title: Medical Treatment Alone Versus Varicocelectomy Versus Varicocelectomy and Medical Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Marwan Mohamed Ali, Resident of Urology, Faculty of Medicine, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Isolated Teratozoospermia
Record Dates: First submitted 2025-05-28; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-09

CONDITIONS: Teratozoospermia
MeSH Terms: conditions — Teratozoospermia | interventions — Carnitine; Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group of l-carnitine and antioxidant (Active Comparator): About 42 male patients suffering from teratozoospermia will take medical treatment (l-carnitine and antioxidant) once daily for 3 months
  Interventions: Drug: l-carnitine
- Group of varicocelectomy (Active Comparator): About 42 male patients suffering from teratozoospermia will undergo subinguinal varicocelectomy.
  Interventions: Drug: l-carnitine
- Group of Mixed Treatment(varicocelectomy then l-carnitine and antioxidant) (Active Comparator): About 42 male patients suffering from teratozoospermia will undergo subinguinal varicocelectomy then adjuvant treatment (l-carnitine and antioxidant) for 3 months.
  Interventions: Drug: l-carnitine

INTERVENTIONS:
Drug: l-carnitine — to compare the efficacy of medical treatment (l-carnitine and antioxidants) versus surgical treatment (varicocelectomy) versus surgical treatment and medical treatment (varicocelectomy with adjuvant medications) on pregnancy rate on varicocele related subfertility patients with isolated teratozoospermia.
  Other Names: Antioxidants; varicocelectomy

SUMMARY:
A varicocele is defined as an abnormal venous dilatation and/or tortuosity of the pampiniform plexus in the scrotum. Although varicoceles are almost always and more common on the left side, up to 50% of the men with varicocele, have bilateral varicoceles.

Varicocele has a negative impact on spermatogenesis, testicular volume, Standard semen parameters, and fertilization, implantation, and embryo outcomes.

DETAILED DESCRIPTION:
Varicocelectomy remains the first-line treatment option in infertile men with palpable varicocele and abnormal semen parameters, with the microsurgical subinguinal approach conveying the greatest success rate and fewest complications. The empirical use of antioxidant supplement may confer some benefits in men to reduce oxidative damage.

Medical management, including antioxidants, could offer a potential solution with lower risks given the increasing evidence suggesting the role of oxidative stress in varicocele-induced infertility.

Physical examination of the scrotum remains the most commonly used technique to diagnose varicoceles. Palpation of the scrotum is best performed in a relaxed patient in standing position, in a warm room and carried out by a well-trained physician.

Surgical treatment of varicocele has a significant effect on semen parameters, so it is considered the 'gold standard' treatment for subfertile males with palpable varicoceles associated with abnormal semen analysis.

ELIGIBILITY:
Inclusion Criteria:

* Sub-fertile men with clinically palpable varicoceles ( unilateral or bilateral ).
* Men with teratozoospermia.

Exclusion Criteria:

* Recurrent varicoceles.
* Significant medical diseases as: Hepatic insufficiency.
* Hypersensitivity to the drugs.
* Female factor of infertility.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment of Teratozoospermia | 3 months
  Treatment of the male patients that suffering from abnormally shaped sperms (Teratozoospermia) by medical treatment and or subinguinal varicocelcetomy

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Sayed Abdel-Kader, Professor, Study Chair — Urology Department, Faculty of Medicine, South Valley University, Qena, Egypt
Locations (1):
- South Valley University Hospital, Qina, South Valley, Egypt

IPD SHARING:
Plan to Share IPD: Undecided